CLINICAL TRIAL: NCT01047813
Title: The Effects of High and Low GI Breakfasts on Cognitive Performance in Adults With Type 2 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leeds (Other)
Responsible Party: Mr Daniel Lamport, Institute of Pscyhological Sciences, University of Leeds
Other Study IDs: 09/H1305/15
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2009-07

CONDITIONS: Type 2 Diabetes
Keywords: Cognitive performance; Type 2 diabetes; Blood glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Type 2 diabetes: This group contains 25 participants with type 2 diabetes
- control group: This group contains 25 participants withput type 2 diabetes. The control group is matched with age, education and lifestyle to the diabetes group.

SUMMARY:
Consumption of a low glycemic index (GI) diet has been shown to improve glycaemic control in type 2 diabetics(Brand-Miller et al., 2003; Jenkins et al., 2008). In addition to the benefits for glycaemic control there is some evidence for acute improvements in cognitive performance after consumption of low GI foods compared with high GI foods in both adults (Benton et al., 2003; Kaplan et al., 2000) and adolescents (Ingwersen et al., 2007; Smith and Foster, 2008).

Given these findings it is possible that low GI focused dietary interventions designed to improve glycaemic control and health outcomes for diabetic patients could also improve the cognitive function of these patients. This is of particular relevance in light of the evidence associating type 2 diabetes with cognitive decrements (Awad et al., 2004; Stewart and Loilitsa 1999; van Harten et al., 2006). To date two studies with type 2 diabetics have reported that a low GI breakfast was associated with increased verbal memory performance compared to a high GI breakfast (Greenwood et al., 2003; Papanikolaou et al. 2006). Further research should investigate the benefit of low GI foods to cognition.

The aim of this study is to examine the effects of high and low glycaemic index breakfast on cognitive performance in adults with type 2 diabetes. Participants will perform a battery of cognitive tests after consuming 3 different breakfasts (high GI, low GI, and water) on 3 different tests days. The participants will be recruited from the general public and from the Leeds Teaching Hospital diabetes clinic.

This research can benefit the development of specific dietary behaviours aimed at reducing diabetes related cognitive decline. This research is part of a PhD funded by the Economic and Social Research Council and the University of Leeds.

DETAILED DESCRIPTION:
The study will conform to a randomised mixed design. Both the diabetic experimental group and the control group will take part in three conditions whereby participants will receive a high GI, a low GI, or a water breakfast delivered in a counterbalanced order. Participants will then perform the battery of cognitive tests on 2 occasions throughout the morning; 30 minutes after breakfast and 180 minutes after breakfast. Blood glucose will be measured from capillary finger-prick blood samples using diabetic glucose meters throughout the morning.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Type 2 diabetes
* White British or White North American ethnicity and native English speakers
* Not previously received or currently received subcutaneous insulin as part of their diabetes treatment.
* Vision sufficiently good to complete the cognitive testing (using glasses and/or lenses).

Exclusion Criteria:

* Dementia (as indicated using the Mini Mental State Examination <26)
* Current (or recent i.e. in last 6 months) cigarette smoker
* Neurological disorder
* Previous stroke
* Medication other than diabetes treatment medication that has a direct effect on the brain and is likely to influence cognitive function.

Co-existent diabetic complications will not be considered exclusion criteria unless they result in inability to complete the cognitive testing (e.g. insufficient vision).

These exclusion criteria have been chosen on the basis that these are factors that can affect cognitive performance. Given that the cognitive tests involve learning English words, only participants who have English as their first language can be included because different cognitive processes are used when learning in a non-native language (Wong et al., 2004). Ethnicity can influence glucose regulation and risk of diabetes. Given that part of this research is examining the relationship between glucose regulation and cognition it is important that potential confounds such as ethnicity/genetic propensity to diabetes are controlled for.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the general population using emails and posters. These will be distributed throughout the University of Leeds, Leeds Metropolitan University, and NHS sites in Leeds. GP's and diabetes specialist doctors and nurses will be asked to inform potential participants of the nature of the study. Ideally spouses, siblings or other close friends/relatives of the experimental group will be recruited for the control group in an attempt to control for education, social class and general lifestyle.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-03 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Cognitive performance (e.g. memory, attention, reaction time, and problem solving ability). | The primary outcome is measured on three occasions during the three conditions
Blood glucose levels | These are measured during of each of the three conditions

SECONDARY OUTCOMES:
Subjective sensations of appetite, mood, and mental alertness | These are measured during all three conditions
Sleep quality | This is measured prior to each of the three test days and at the screening visit
Stress levels | This is measured prior to each of the three test days and at the screening visit

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Psychological Sciences, University of Leeds, UK, Leeds, West Yorkshire, United Kingdom

REFERENCES:
- [Background] Awad N, Gagnon M, Messier C. The relationship between impaired glucose tolerance, type 2 diabetes, and cognitive function. J Clin Exp Neuropsychol. 2004 Nov;26(8):1044-80. doi: 10.1080/13803390490514875. PMID 15590460
- [Background] Benton D, Ruffin MP, Lassel T, Nabb S, Messaoudi M, Vinoy S, Desor D, Lang V. The delivery rate of dietary carbohydrates affects cognitive performance in both rats and humans. Psychopharmacology (Berl). 2003 Feb;166(1):86-90. doi: 10.1007/s00213-002-1334-5. Epub 2002 Dec 12. PMID 12488949
- [Background] Brand-Miller J, Hayne S, Petocz P, Colagiuri S. Low-glycemic index diets in the management of diabetes: a meta-analysis of randomized controlled trials. Diabetes Care. 2003 Aug;26(8):2261-7. doi: 10.2337/diacare.26.8.2261. PMID 12882846
- [Background] Greenwood CE, Kaplan RJ, Hebblethwaite S, Jenkins DJ. Carbohydrate-induced memory impairment in adults with type 2 diabetes. Diabetes Care. 2003 Jul;26(7):1961-6. doi: 10.2337/diacare.26.7.1961. PMID 12832296
- [Background] Ingwersen J, Defeyter MA, Kennedy DO, Wesnes KA, Scholey AB. A low glycaemic index breakfast cereal preferentially prevents children's cognitive performance from declining throughout the morning. Appetite. 2007 Jul;49(1):240-4. doi: 10.1016/j.appet.2006.06.009. Epub 2007 Jan 16. PMID 17224202
- [Background] Jenkins DJ, Kendall CW, McKeown-Eyssen G, Josse RG, Silverberg J, Booth GL, Vidgen E, Josse AR, Nguyen TH, Corrigan S, Banach MS, Ares S, Mitchell S, Emam A, Augustin LS, Parker TL, Leiter LA. Effect of a low-glycemic index or a high-cereal fiber diet on type 2 diabetes: a randomized trial. JAMA. 2008 Dec 17;300(23):2742-53. doi: 10.1001/jama.2008.808. PMID 19088352
- [Background] Kaplan RJ, Greenwood CE, Winocur G, Wolever TM. Cognitive performance is associated with glucose regulation in healthy elderly persons and can be enhanced with glucose and dietary carbohydrates. Am J Clin Nutr. 2000 Sep;72(3):825-36. doi: 10.1093/ajcn/72.3.825. PMID 10966906
- [Background] Papanikolaou Y, Palmer H, Binns MA, Jenkins DJ, Greenwood CE. Better cognitive performance following a low-glycaemic-index compared with a high-glycaemic-index carbohydrate meal in adults with type 2 diabetes. Diabetologia. 2006 May;49(5):855-62. doi: 10.1007/s00125-006-0183-x. Epub 2006 Mar 1. PMID 16508776
- [Background] Smith MA, Foster JK. The impact of a high versus a low glycaemic index breakfast cereal meal on verbal episodic memory in healthy adolescents. Nutr Neurosci. 2008 Oct;11(5):219-27. doi: 10.1179/147683008X344110. PMID 18782482
- [Background] Stewart R, Liolitsa D. Type 2 diabetes mellitus, cognitive impairment and dementia. Diabet Med. 1999 Feb;16(2):93-112. doi: 10.1046/j.1464-5491.1999.00027.x. PMID 10229302
- [Background] van Harten B, de Leeuw FE, Weinstein HC, Scheltens P, Biessels GJ. Brain imaging in patients with diabetes: a systematic review. Diabetes Care. 2006 Nov;29(11):2539-48. doi: 10.2337/dc06-1637. No abstract available. PMID 17065699
- [Background] Wong PC, Parsons LM, Martinez M, Diehl RL. The role of the insular cortex in pitch pattern perception: the effect of linguistic contexts. J Neurosci. 2004 Oct 13;24(41):9153-60. doi: 10.1523/JNEUROSCI.2225-04.2004. PMID 15483134
- [Derived] Lamport DJ, Dye L, Mansfield MW, Lawton CL. Acute glycaemic load breakfast manipulations do not attenuate cognitive impairments in adults with type 2 diabetes. Clin Nutr. 2013 Apr;32(2):265-72. doi: 10.1016/j.clnu.2012.07.008. Epub 2012 Aug 15. PMID 22959621